CLINICAL TRIAL: NCT07049705
Title: Factors Influencing Bradycardia During Spinal Anesthesia in Obstetric Patients Undergoing Cesarean Section
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/916
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study titled "Factors Influencing Bradycardia During Spinal Anaesthesia in Obstetric Patients Undergoing Caesarean Section"" aims to investigate the causes and patterns of bradycardia in pregnant women receiving spinal anesthesia during cesarean deliveries. Bradycardia, defined as a heart rate below 60 beats per minute, is a known complication of spinal anesthesia, often resulting from sympathetic blockade and unopposed parasympathetic activity. This condition may lead to hypotension, decreased cardiac output, and compromised fetal oxygenation.

DETAILED DESCRIPTION:
The research seeks to enhance the understanding of both patient-specific and procedural risk factors, contributing to improved clinical management, safer anesthesia practices, and better maternal-fetal outcomes. Ethical approval and informed consent protocols are included to ensure participant safety and data confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients aged 18-40 years.
* Undergoing elective or emergency cesarean sections under spinal anesthesia.
* Classified as ASA Physical Status I or II (relatively healthy or with mild systemic disease).
* Provided informed consent (either by the patient or legal guardian).

Exclusion Criteria:

* Patients with pre-existing cardiac conditions (e.g., arrhythmias, conduction abnormalities).
* Patients taking medications that affect heart rate, such as beta-blockers or calcium channel blockers.
* Patients with contraindications to spinal anesthesia (e.g., coagulopathy, infection at the injection site).
* Those undergoing combined spinal-epidural or general anesthesia.
* Patients with incomplete medical records or unable to provide informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The research seeks to enhance the understanding of both patient-specific and procedural risk factors, contributing to improved clinical management, safer anesthesia practices, and better maternal-fetal outcomes. Ethical approval and informed consent protocols are included to ensure participant safety and data confidentiality.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
structured questionnaire | 12 Months
  1. Section A: Demographic and Baseline Information
     Age, weight, height, gestational age, parity, medical history, medications.
  2. Section B: Anesthetic and Surgical Details
     Indication for cesarean (elective/emergency), baseline heart rate and BP, type/dose of anesthetic, sensory block level, fluid administration, blood loss.
  3. Section C: Intraoperative Hemodynamic Events
     Occurrence of bradycardia (HR < 60 bpm), lowest HR, time to bradycardia, associated hypotension, interventions used, maternal symptoms.
  4. Section D: Neonatal Outcomes
  Apgar scores at 1 and 5 minutes, NICU admission and reasons.
  Scoring:
  There is no numerical scoring system described. Instead:
  Responses are mostly categorical or numerical entries (e.g., Yes/No, HR value, BP value, Apgar score).

CONTACTS AND LOCATIONS:
Locations (1):
- Maqsood Medical complex, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No